CLINICAL TRIAL: NCT01611259
Title: Phase II Trial of Rituximab Plus Lenalidomide in Patients With Lymphoma of the Mucosa Associated Lymphoid Tissue (MALT) Type
Brief Title: Rituximab Plus Lenalidomide in Patients With Mucosa Associated Lymphoid Tissue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_MALT2
Record Dates: First submitted 2012-05-18; First posted 2012-06-04 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-06

CONDITIONS: Lymphoma of the Mucosa Associated Lymphoid Tissue (MALT)
Keywords: MALT Lymphoma; Lenalidomide; Rituximab; AGMT
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab and Lenalidomide (Experimental): Single arm: 6 cycles for patients with complete response, 8 cycles for subjects with stable disease or partial remission; cycles duration: 28 days Rituximab (Mabthera®): 375 mg/m² i.v. day 1 Lenalidomide (Revlimid®): 20 mg p.o. daily for 21 days
  Interventions: Drug: Rituximab and Lenalidomide

INTERVENTIONS:
Drug: Rituximab and Lenalidomide — Rituximab 375 mg/m² i.v. day 1 Lenalidomide 20 mg p.o. daily for 21 days Cycles should be repeated every 28 days. Restaging should be performed after three cycles. In case of at least stable disease, patients should receive another three courses of therapy. Patients with documented CR after 6 courses will stop therapy/study, while patients with PR or SD will be given another two cycles for a maximum of 8 cycles.

SUMMARY:
This is an open label, phase II study to evaluate the capacity of Rituximab (Mabthera®) plus Lenalidomide (Revlimid®) to induce objective responses in patients with Mucosa Associated Lymphoid Tissue (MALT) lymphoma presenting with measurable disease.

ELIGIBILITY:
Inclusion Criteria selected:

* Histologically verified diagnosis if MALT lymphoma of any localization
* Measurable disease upon diagnosis or first or greater relapse after local therapy, prior chemotherapy orHP-eradication. In addition, also in patients with gastric MALT-lymphoma judged refractory to HP-eradication by a minimum follow-up of 12 months after successfulHP-eradication will be included in the study. Patients with gastric MALT lymphoma and no evidence of HP-infection may be enrolled immediately
* Ann Arbor Stage I-IV
* In case of prior treatment with Rituximab, the presence of CD20 on lymphoma cells must have been demonstrated before inclusion in the trial.
* ECOG performance status of 0,1 or 2
* Patient must be able to take aspirin daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin

Exclusion Criteria selected:

* Lymphoma histology other than MALT lymphoma or MALT lymphoma with a diffuse large cell lymphoma ("high grade lymphoma") - component
* Use of any investigational agent within 28 days prior to initiation of treatment with lenalidomide
* History of malignancy other than squamous cell carcinoma, basal cell carcinoma of the skin or carcinoma in situ of the cervix within the last 5 years
* Major surgery, other than diagnostic surgery, within the last 4 weeks
* Evidence of CNS involvement
* A history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and adversely affecting compliance to study drugs
* Severe peripheral polyneuropathy
* Clinically significant cardiac disease or myocardial infarction within the last 6 months
* Known hypersensitivity to thalidomide or lenalidomide or rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Raderer, MD, Principal Investigator — Allgemeines Krankenhaus der Stadt Wien - Medizinischer Universitätscampus
Locations (5):
- Austria (5):
  - AKH Linz, Linz, Upper Austria
  - Klin.Abt.f. Hämatologie; Med.Univ.Graz, Graz
  - Univ.-Klinik f. Innere Medizin V, Innsbruck
  - PMU Salzburg, Salzburg
  - Universitätsklinik f. Innere Medizin I, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kiesewetter B, Willenbacher E, Willenbacher W, Egle A, Neumeister P, Voskova D, Mayerhoefer ME, Simonitsch-Klupp I, Melchardt T, Greil R, Raderer M; AGMT Investigators. A phase 2 study of rituximab plus lenalidomide for mucosa-associated lymphoid tissue lymphoma. Blood. 2017 Jan 19;129(3):383-385. doi: 10.1182/blood-2016-06-720599. Epub 2016 Nov 22. No abstract available. PMID 27879257
- See also: Sponsor — http://www.agmt.at

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 50 patients were enrolled at 4 sites in Austria. First patient in was 06-Jun-2012; Last patient in was 26-May-2014.
Pre-assignment Details: 2 patients were withdrawn before first response evaluation and were replaced. 2 patients withdrew their consents prior to study treatment and did not experience AEs to other study procedures. These 2 patients were therefore excluded from intent-to-treat (ITT) efficacy assessments, safety assessments and listing of baseline characteristics.
Groups:
- Rituximab and Lenalidomide: Rituximab was administered on day 1 of each cycle in a dose of 375 mg/m² (28 day cycle). Dose of lenalidomide for investigation is 20 mg/day, orally on days 1 to 21 followed by 7 days pause.Restaging should be performed after three cycles. In case of at least stable disease, patients should receive another three courses of therapy. Patients with documented CR after 6 courses stopped therapy/study, while patients with PR or SD were given another two cycles for a maximum of 8 cycles.
Period: Overall Study
Arm/Group | Rituximab and Lenalidomide
Started | 48
Completed | 34
Not Completed | 14
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Population: Two of the enrolled patients withdrew their consent prior to study treatment and did not experience adverse events due to other study procedures. These 2 patients were therefore excluded from intent-to-treat (ITT) and per-protocol (PP) efficacy assessments, safety assessments and listing of baseline characteristics.
Arm/Group | Rituximab and Lenalidomide
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 65 [33 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Objective Responses in Patients With MALT Lymphoma Presenting With Measureable Disease
Description: The primary objective of this Phase II study is to evaluate the proportion of patients responding to Lenalidomide and Rituximab. In case of a response rate of < 40%, the combination is rejected as ineffective, while an active combination is defined at a minimum response rate of 60% based of findings with rituximab and lenalidomide mono-therapy.
Time Frame: 40 weeks
Population: 48 patients were included into safety assessment, two of them received treatment but no efficacy assessment was available. Therefore, these two patients were neither included into Intention-to-treat nor Per-protocol efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab and Lenalidomide
Number analyzed (Participants) | 46
Participants
  CR | 25
  PR or SD | 20
  PD | 1

2. Secondary Outcome: Number and Severity of Adverse Events
Description: Safety of Rituximab (Mabthera®) plus Lenalidomide (Revlimid®) in this patient population
Time Frame: From treatment start until 28 days after last study treatment; expected study duration 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Influence of Rituximab Plus Lenalidomide on T-cell Subsets
Description: T-cell subsets will be evaluated from EDTA blood in a central lab
Time Frame: Day 1, 14 and 28 of cycle 1 and day 1 of cycle 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All AEs were recorded by the Investigator from the time the subject signs informed consent to 28 days after the last dose of study medication.
Arm/Group | Rituximab and Lenalidomide
Serious Adverse Events (participants affected / at risk) | 18/48
Other Adverse Events (participants affected / at risk) | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab and Lenalidomide (N=48)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Colecystitis (Hepatobiliary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.17% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab and Lenalidomide (N=48)
Leucocyte count (Blood and lymphatic system disorders) | 6 (15)
Conjunctivitis (Eye disorders) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 9 (16)
Dry mouth (Gastrointestinal disorders) | 4 (5)
Dysgeusia (Gastrointestinal disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (4)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 3 (3)
Meteorism (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (10)
Stomatitis (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 5 (5)
Chills (General disorders) | 9 (10)
Condition aggravated (General disorders) | 2 (2)
Fatigue (General disorders) | 17 (20)
Infusion related reaction (General disorders) | 2 (4)
Mucositis (General disorders) | 2 (3)
Night sweats (General disorders) | 3 (4)
Oedema peripheral (General disorders) | 5 (6)
Pyrexia (General disorders) | 8 (9)
Hypersensitivity (Immune system disorders) | 5 (6)
Bronchitis (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2)
Oral herpes (Infections and infestations) | 4 (4)
Overdose (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Haemoglobin (Investigations) | 3 (5)
Lymphocyte count (Investigations) | 3 (6)
Neutrophil count (Investigations) | 12 (28)
Platelet count (Investigations) | 3 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (15)
Headache (Nervous system disorders) | 6 (11)
Insomnia (Nervous system disorders) | 5 (6)
Tremor (Nervous system disorders) | 2 (3)
Vertigo (Nervous system disorders) | 11 (12)
Nocturia (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Eyelid oedema (Skin and subcutaneous tissue disorders) | 2 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (34)
Rash (Skin and subcutaneous tissue disorders) | 23 (39)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other